CLINICAL TRIAL: NCT00299273
Title: Exploratory Feasibility Study: High Fat/Protein Diet in the Treatment of Obesity
Brief Title: High Fat - High Protein Diet in the Treatment of Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Rockefeller University (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JBR-0583; NCT00503373 (obsolete NCT alias)
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: Obesity;; Low calorie high fat/protein diet;; Low-carbohydrate diet; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low calorie high fat/protein diet (Experimental): Low calorie high fat/protein diet
  Interventions: Behavioral: Low calorie high fat/protein diet

INTERVENTIONS:
Behavioral: Low calorie high fat/protein diet — 6 weeks of caloric restriction (50%) on a high fat/protein diet

SUMMARY:
The purpose of this study is to examine the effects of a low calorie high fat/protein diet on body fat and body composition in overweight and obese subjects. The investigators will also test the effects of this diet on secondary outcomes such as: fluid and electrolyte balance, cholesterol, inflammation, sugar and insulin metabolism, fat hormones, blood pressure and feelings of fullness.

DETAILED DESCRIPTION:
Participation in this study requires 2 screening visits to the outpatient clinic, and if participants qualify, 10 inpatient study weeks.

Subjects will be admitted to the Rockefeller University Hospital for the 10 week in-patient phase of the study. The first 2 weeks consist of a weight stabilization period, during which subjects will be required to eat an average American diet. This is followed by the 6 week weight loss period where subjects will be put on a low calorie high fat/protein diet. During the weight loss period, calories will be cut by 50% compared to the weight stabilization period. This will be followed by a 2 week weight maintenance period during which calories will be added to the diet to maintain the new weight. Appropriate adjustments will be made to keep the subject's weight stable.

During the entire inpatient study, subjects will consume one multivitamin per day (Centrum, always complete, from A to Zinc) and one iron supplement per day. In addition, unlimited access to zero calorie liquids (water/diet soda) will be available and subjects will be encouraged to maintain their usual activity level.

Females of reproductive age need to make sure that they do not become pregnant during the inpatient study. Urine will be tested for pregnancy once during each phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 30 to 34.9 or
* BMI of 25 to 29.9 and a waist circumference > 88cm (35in)
* Pre-menopausal-

Exclusion Criteria:

* High Blood Pressure
* High Cholesterol
* Diabetes
* Anemia
* Liver disease
* Kidney disease
* HIV positive
* Syphilis
* Hepatitis B/C positive

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2006-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Visceral adipose tissue | after 6 weeks

SECONDARY OUTCOMES:
Body composition, fluid and electrolyte balance, lipids/lipoprotein metabolism, markers of inflammation, glucose and insulin metabolism, fat hormones, blood pressure and measures of satiety. | after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan L. Breslow, MD, Principal Investigator — The Rockefeller University Hospital
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States